CLINICAL TRIAL: NCT03344848
Title: Early Feasibility Study of the Orion Visual Cortical Prosthesis System
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Sight Medical Products (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CP-07; 5UH3NS103442 (NIH)
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Blindness, Acquired
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single Arm (Experimental): Implanted with the Orion Visual Cortical Prosthesis System
  Interventions: Device: Orion Visual Cortical Prosthesis System

INTERVENTIONS:
Device: Orion Visual Cortical Prosthesis System — The Orion Visual Cortical Prosthesis System is intended to stimulate the medial surface of the occipital lobe in the visual cortex to induce visual perception in blind individuals.

SUMMARY:
This is an early feasibility study of a new device, the Orion Visual Cortical Prosthesis System. The device is intended to stimulate the surface of the visual cortex to induce visual perception in blind individuals.

DETAILED DESCRIPTION:
In this study, 6 subjects with bare light or no light perception in both eyes will be implanted with the Orion Cortical Visual Prosthesis System. The study will evaluate the safety of the device and surgery, as well as reliability of the system and the usefulness of any restored vision. Each subject will be followed for 6 years, with their health monitored throughout. Research sessions, visual function testing, and subject-reported outcomes will be used to evaluate the functioning of the system.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is bilaterally blind with bare or no light perception. This is defined as non-measurable binocular visual acuity or 5° or less visual field in each eye.
2. Subject is bilaterally blind due to:

   1. Trauma to the eye, or
   2. Disease or damage of the retina (such as retinopathy, retinal vein occlusion, inherited retinal diseases or retinal detachment), or
   3. Disease or damage of the optic nerve or chiasm (such as glaucoma, methanol intoxication, autoimmune neuropathies, pituitary pathology, and hereditary neuropathies)
3. Subject's vision cannot be restored with any approved medication or intervention.
4. Subject has a documented history of useful form vision.
5. Subject is between the age of 22-74 .
6. Subject resides within 2 hours (by ground transportation) of the investigational site.
7. Subject is (a) male or (b) a female of childbearing potential with a negative pregnancy test who is using a reliable method of contraception or (c) a female who is at least two years post-menopause or otherwise unable to bear children.
8. Subject is able to complete regular office and telephone appointments per the protocol requirements.
9. Subject is medically fit for neurosurgical intervention.

Exclusion Criteria:

1. Subject is at high risk for surgical complications such as active systemic infection, coagulation disorders (such as the use of anti-thrombotic therapies) or platelet count below 100,000.
2. Subject has history of bleeding or immune compromise.
3. Subject is taking chronic anticoagulants or antiplatelet agent or subject has an abnormally elevated preoperative coagulation profile (either PTT or PT/INR).
4. Subject has had prior craniotomy or brain surgery that would interfere with placement or function of Orion device.
5. Subject has evidence of active intracranial disease that would preclude elective neurosurgical intervention, such as unruptured intracranial aneurysm or brain tumor, or aberrant visual cortex anatomy, such as prior stroke or arteriovenous malformation.
6. Subject has a significant abnormality on preoperative brain MRI.
7. Subject has a prior history of seizures or epilepsy.
8. Subject has Parkinson's disease.
9. Subject has a prior history of serious head injury with loss of consciousness for more than 24 hours.
10. Subject has a progressive central nervous system disease.
11. Subject has a history of implant-related infection.
12. Subject requires or is likely to require any of the following medical procedures while implanted with the Orion System: MR imaging, diathermy, electroconvulsive therapy (ECT), or transcranial magnetic stimulation (TMS). These medical procedures are contraindicated for subjects implanted with an Orion System. Energy from these procedures can be sent through the implanted brain stimulation system and cause permanent brain damage which may cause severe injury, coma, or death.
13. Subject is implanted with any neurostimulation or neuromodulation device in the head including, but not limited to cochlear implant, deep brain stimulator, or auditory brain implant.
14. Subject has a clinically significant or unstable medical condition including uncontrolled systemic hypertension with values above 170/100; cardiac or pulmonary disease; uncorrected coagulation abnormalities; diabetes; or any condition that would render the patient unable to safely cooperate with the study tests as judged by the screening physician.
15. Subject has had an alcohol or illicit substance use disorder within the last 6 months, unstable remission of substance abuse, or chart evidence that co-morbid substance use disorder could account for lack of treatment response.
16. Subject has uncontrolled chronic pain.
17. Subject has significant neurocognitive impairment in memory domain (based on MoCA-BLIND <18 or WAIS-IV <80, described below).
18. Subject had moderate or severe depression, as determined by a score of at least 17 on the HAM-D.
19. Subject has had a suicide attempt in the last two years, presence of a suicide plan (an answer of "Yes" to Question C4 in Section C-Suicidality of MINI International Neuropsychiatric Interview), or a "yes" answer to any one of the ten suicidal ideation and behavior questions on the C-SSRS.
20. Subject has a disease or condition that prevents understanding or communication of informed consent, study demands, or testing protocols, including:

    1. Cognitive decline including diagnosed forms of dementia and/or progressive neurologic disease
    2. Psychiatric disease including diagnosed forms of depression
    3. Does not speak a principal language associated with the region
    4. Deafness or selective frequency hearing loss that prevents adequate communication with the researchers.
21. Subject has a balance disability or frequently participates in contact sports.
22. Subject must administer diathermy as part of his/her livelihood.
23. Subject is pregnant or is planning on becoming pregnant in the next year.
24. Subject has unrealistic expectations of the benefits of the study.
25. Subject is enrolled in another therapeutic investigational drug or device trial

Ages: 22 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of Device- or Procedure-Related Adverse Events (Safety) | Through study completion, an average of 6 years
  Collection of adverse events

SECONDARY OUTCOMES:
Ability to Create Visual Perception as Measured by Stimulation Thresholds | 1 month, 6 months, 12 months, 24 months, 60 months, 72 months
  Measurement of stimulation thresholds on each electrode or groups of electrodes

CONTACTS AND LOCATIONS:
Overall Officials: Uday Patel, PhD, Study Director — Second Sight Medical Products
Locations (2):
- United States (2):
  - University of California, Los Angeles, Los Angeles, California
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beauchamp MS, Oswalt D, Sun P, Foster BL, Magnotti JF, Niketeghad S, Pouratian N, Bosking WH, Yoshor D. Dynamic Stimulation of Visual Cortex Produces Form Vision in Sighted and Blind Humans. Cell. 2020 May 14;181(4):774-783.e5. doi: 10.1016/j.cell.2020.04.033. PMID 32413298